CLINICAL TRIAL: NCT07109570
Title: Surface Electrical Myography, Oxygen Consumption (VO2), Effort, and Weaning in the Mechanically Ventilated Patient in the Intensive Care Unit (ICU): SERA-Effort Study
Brief Title: Surface Electrical Myography, Oxygen Consumption, Effort, and Weaning in the Mechanically Ventilated Patient in the Intensive Care Unit
Acronym: SERA-Effort
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Demcon-Macawi (Unknown)
Responsible Party: Principal Investigator, Abraham Schoe, MD, PhD., MD, PhD, Leiden University Medical Center
Other Study IDs: P24.116; NL86876.058.24 (Other: ToetsingOnline)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Intensive Care Units (ICUs); Weaning Failure; Mechanical Ventilation; Spontaneous Breathing Trial; Diaphragm Electrical Activity; Oxygen Consumption
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to measure effort using esophageal pressure measurements, oxygen consumption and diaphragm activity in mechanically ventilated Intensive Care Unit patients during a Spontaneous Breathing Trial. The main question aims to answer whether the sEMG signal derived from the SERA device, effort parameters and oxygen consumption have an association with weaning failure.

Participants will be measured while performing a spontaneous breathing trial.

DETAILED DESCRIPTION:
Rationale: In patients mechanically ventilated for more than 72 hours weaning from the ventilator and successful extubation can be problematic. The spontaneous breathing trial (SBT) is a tool to predict successful extubation. However re-intubation withing 48 hours occurs in 15-20% of the patients after a successful SBT. The key parameter of the SBT is the rapid shallow breathing index (RSBI). Since the rate of extubation failure is still high the search for a better parameter than the RSBI is warranted.

Recently measurement of the surface electromyography of the respiratory muscles has become available with the Surface Electromyography Respiratory Assist (SERA), which has been developed by Demcon-Macawi. The device is currently investigated in neonates in search of an apnea detection algorithm (protocol ID NL83937.000.23). The device gives an estimate of the magnitude of the electric activity of the diaphragm which has a good correlation with the force the diaphragm generates. It is known that the diaphragm is the key respiratory muscle and that dysfunction of the diaphragm has a strong association with weaning failure. We think that this signal could be of great value in detecting weaning and extubation failure therefore we want to investigate if the sEMG signal derived from the SERA device has an association with weaning failure, defined as an unsuccessful SBT, or extubation failure, defined as the need for re-intubation for respiratory reasons within 48 hours after a successful SBT and subsequent extubation.

Objective: Primary objective is to investigate if the sEMG signal derived from the SERA device has an association with weaning failure, defined as an unsuccessful SBT, or extubation failure, defined as the need for re-intubation for respiratory reasons within 48 hours after a successful SBT and subsequent extubation.

Secondary objectives are to investigate if the sEMG signal has an association with other measurements of effort (pressure time product (PTP), Work of breathing (WOB), Transpulmonary pressure swings, oesophageal pressure swings, and oxygen consumption).

Study design: A single center prospective cohort feasibility/pilot study performed on patients undergoing a spontaneous breathing trial. Measurements will commence 10 minutes before the planned SBT, will continue during the SBT until 10 minutes after the termination of the SBT. Measurement data will be derived from the SERA, the mechanical ventilator (Hamilton C6), and the Masimo ISA OR+. The SBT will done according to the ruling protocol in the LUMC.

Intervention: None Main study parameters/endpoints: Magnitude of the electric signal (base level, or tonic level, maximum level, AUC of the electric signal during contraction in inspiration and expiration, differences between maximum and tonic levels), VO2, PTP, WOB, RSBI, diaphragmatic pressure swing.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: The collection of data will not affect the standard of care. Therefore, the patient's risk is negligible and the burden is minimal.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Esophageal catheter in situ (standard of care)
* Eligible for an SBT in the near future according to the LUMC SBT protocol currently valid

Exclusion Criteria:

* Severe cardiac failure NYHA class IV without mechanical support (LVAD or Impella)
* COPD Gold IV
* Pregnancy
* Patients with ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population consists of adults who are mechanically ventilated in the ICU and meet the criteria for a regular spontaneous breathing trial according to the ruling LUMC protocol.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | 48 hours after extubation
  Extubation failure is defined by the need for reintubation or death.
sEMG differences during SBT | 10 minutes before switch from support to no support ventilation, the whole duration of the SBT, and the 10 minutes after the SBT when there is again support.
  The AUC of the voltage signal, the phasic level (difference between tonic level and maximum level) and the tonic level (base level).

SECONDARY OUTCOMES:
Differences of oxygen consumption during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of oxygen consumption (in milliliter/minute) and the differences between start, during, and end of the SBT.
Differences of esophageal pressure swings measured with an esophageal catheter during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of pressure swings (in cmH2O), measured with an esophageal catheter, and the differences between start, during, and end of the SBT.
Differences of work of breathing measured with an esophageal catheter during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of work of breathing (in Joules/liter), measured with an esophageal catheter, and the differences between start, during, and end of the SBT.
Differences of pressure-time product measured with an esophageal catheter during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of pressure-time product (in cmH2O/seconds), measured with an esophageal catheter, and the differences between start, during, and end of the SBT.
Differences of rapid shallow breathing index during SBT | 10 minutes before, through SBT (average of 30 minutes) and 10 minutes after SBT
  The values of rapid shallow breathing index (breaths/minute/liter) and the differences between start, during, and end of the SBT.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Centre, Leiden, Netherlands